CLINICAL TRIAL: NCT03418896
Title: Novel Extragonadal Effects of Human Chorion Gonadotropin (hCG) on Calcium Homeostasis
Brief Title: Extragonadal Effects of hCG on Calcium Homeostasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Martin Blomberg Jensen (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, Group leader, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-003546-84
Record Dates: First submitted 2018-01-05; First posted 2018-02-01 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hypogonadism; Calcium Disorder; Renal Disease
MeSH Terms: conditions — Hypogonadism; Kidney Diseases | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Intervention Model Description: simple one arm intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- human chorion gonadotropin (Experimental): Pregnyl, hCG, 5000 IU times one im.
  Interventions: Drug: human chorionic gonadotropin

INTERVENTIONS:
Drug: human chorionic gonadotropin — a single injection of a standard dose

SUMMARY:
A pilot study showed that serum calcium levels and calcium homeostasis change in response to hCG stimulation test. Serum calcium level differed when comparing pretreatment values at baseline with serum levels 72 hours after hCG stimulation in men with gonadal insufficiency referred for this stimulation test. Now we want to investigate whether this change in calcium is due to renal loss or other mechanisms and how the classical regulators of calcium homeostasis respond to hCG in men with impaired gonadal function compared with men having normal gonadal function. Moreover, the observed change in serum calcium implies that hCG also changes Phosphate, PTH and calcitonin and this will be clarified with this study

DETAILED DESCRIPTION:
Aim To investigate whether human chorionic gonadotropin (hCG) stimulation test changes calcium-phosphate homeostasis in men with normal and impaired testicular function.

The overall purpose of the project is to investigate the importance of human chorion gonadotropin (hCG) for the calcium balance in normal men and men with impaired testicular function.

BACKGROUND AND HYPOTHESES

The Department for Growth and Reproduction has helped to uncover the rising occurrence of early puberty, infertility, polycystic ovarian syndrome and testicular cancer that is worryingly high in large numbers parts of the world (1). These conditions are all governed by the hormonal axis that contains hypothalamus, pituitary gland, and the HPG axis (2). Our hypothesis is, that hCG may be a new regulator of calcium balance. hCG acts like luteinizing hormone (LH) produced by the pituitary gland and stimulates by binding to the LH receptor (LHCGR) production of testosterone in the testicles (3-6). we and others have found that that LHCGR is also located in other tissues than the gonad (7) and we suggest that LH stimulation probably also regulates calcium handling in the kidney. We have observed changes in serum calcium after hCG injection in patients with impaired testicular function, which indicates that the gonads and gonadotropins may be important for calcium and phosphate homeostasis. It is compatible with the fact that it has been shown that ex FSH can regulate bone function (8),and sex hormones are important for calcium absorption and excretion in the kidney (9-11). The latter is interesting because our research suggests that the receptor for the luteinizing hormone and hCG (LHCGR) plays an important role in the kidney, thus enabling a direct effect on calcium and phosphate handling for LHCGR agonists such as LH and hCG.

With this study we want to investigate how hCG influences calcium homeostasis and subsequently other extragonadal organs by analyzing serum and urine from men with normal and impaired gonadal function

DESIGN This is a prospective intervention study in cases and controls

Patients and methods 10-15 men referred for hCG stimulation test due to suspected gonadal insufficiency after curative treatment for testicular cancer with orchiectomy, irradiation or chemotherapy age 18-80 years at Department of growth and reproduction, Rigshospitalet and 10-15 men with normal reproductive function

SAMPLE SIZE CALCULATION AND STATISTICS By using a test level of 5% (level of significance), power of 80% and at least 10 normal men and 10 men with impaired gonadal function completing the trial will enable us to detect a change in serum calcium of 6%, PTH of 25% and a change in serum Phosphate of 15%.

SCREENING AND TIME COURSE Men referred for hCG stimulation test at our Department will be screened for eligibility to the study. Those who meet the criteria for participation will be informed, and if they consent allocated to the study.

Each person will have one blood sampling performed.Venus blood is drawn before hCG administration, 2,8,24 72 and 120 hours after injection. Spot urine samples will be delivered and ECG monitoring will be performed at all time points. All men will be fasting for baseline, 2 hours, 24, 72 and 120 hours sampling. Serum will be send for analysis within 40 minutes and the rest frozen within 1 hour and will be stored at minus 80 degrees celsius until analysis.

Biostatistical analysis each individual's samples will be normalized by division of the value of the given parameter (for instance calcium or phosphate) to the baseline samples drawn before the intervention.

Hence, samples from each volunteer at the different timepoints will be normalized with the individual's own baseline values before the administration of hCG. Initially, paired Student t tests will be used to compare changes in serum or urine by comparing baseline levels with the different time points. Unpaired Student t tests will be used to compare controls and men with gonadal insufficiency at all time points. Moreover, the presumable effect of multiple testing will be tested afterwards by using ANOVA followed by a post hoc Dunnett's /SIDAK multiple comparison test. All data will after indexation to baseline levels be shown as mean ± SEM. Differences were considered statistically significant when P ≤ 0.05.

Predefined subgroups Changes in calcium and phosphate will be analyzed according to baseline sex steroids and delta sex steroids, LHCGR, BMI, GFR, PTH

Principal Investigator: Li Juel Mortensen Sponsor: Martin Blomberg Jensen

ELIGIBILITY:
Inclusion Criteria: to be either

* a man with normal reproductive function
* or a man with known impaired gonadal function
* more than 18 years of age and less than 80 years of age

Exclusion Criteria:

* presence of current serious diseases
* or presence of disease requiring constant and lifelong treatment with chemotherapy or other toxic drugs
* Men treated with testosterone who do not stop their treatment while being part of the study,

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — males
Enrollment: 12 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Serum calcium | 2,8,24, 72,120 hours
  changes albumin corrected calcium, ionized calcium, total calcium

SECONDARY OUTCOMES:
urinary calcium and phosphate excretion | 2,8,24, 72,120 hours
  calcium and phosphate clearance and fractional excretion
serum Phosphate | 2,8,24, 72,120 hours
  changes in serum phosphate

OTHER OUTCOMES:
vitamin D metabolites | 2,8,24, 72,120 hours
  25OHD, 1,25OH2D3, 24,25OH2D3
calcitonin | 2,8,24, 72,120 hours
  changes in serum calcitonin
Cortisol | 2,8,24, 72,120 hours
  Changes in serum cortisol
adrenal steroidogenesis | 2,8,24, 72,120 hours
  all measurable steroids part of steroidogenesis by LCMS
sex steroids | 2,8,24, 72,120 hours
  total and free calculated levels of sex steroids including T/LH
reproductive hormones | 2,8,24, 72,120 hours
  AMH, Inhibin B, FSH, including InhB/FSH
change in adipocyte function | 2,8,24, 72,120 hours
  biomarkers in serum of adipocyte function, browning, differentiation, insulin, glucose, HB1AC etc
LHCGR | 2,8,24, 72,120 hours
  serum LHCGR may change
regulators of calcium homeostasis | 2,8,24, 72,120 hours
  serum calcitonin, FGF23, interferons, prostaglandins
Kidney function | 2,8,24, 72,120 hours
  changes in GFR, creatinine, Urea, pH, HCO3
Electrocardiogram | 2,8,24,72,120 hours
  changes in QT, corrected QY or QRS
adipocyte function | 2,8,24,72,120 hours
  changes in serum lipid or cholesterol or adipocyte function markers
liver function | 2,8,24,72,120 hours
  changes in albumin and hepatic binding proteins
bone function | 2,8,24,72,120 hours
  changes in bone markers such as CTX, osteocalcin and endocrine bone factors RANKL, OPG, RANK, sclerostin
serum PTH | 2,8,24,72,120 hours
  changes in serum PTH
urinary excretion of steroids | 2,8,24,72,120 hours
  cortisol and sex steroids
Cardiovascular biomarkers | 2,8,24,72,120 hours
  ANP and BNP
glucose homeostasis | 2,8,24,72,120 hours
  insulin, glucose, c-peptid, HB1AC, HOMA, Quicki
incretin hormones | 2,8,24,72,120 hours
  glucagon, and GLP-1
electrolytes | 2,8,24,72,120 hours
  Magnesium, potassium, sodium

CONTACTS AND LOCATIONS:
Overall Officials: Martin blomberg Jensen, Study Chair — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Department of Growth and Reproduction, Rigshospitalet, Copenhagen
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided
Normally we share the data through an official danish Databank handling all these things

REFERENCES:
- [Derived] Juel Mortensen L, Lorenzen M, Jorgensen A, Albrethsen J, Jorgensen N, Moller S, Andersson AM, Juul A, Blomberg Jensen M. Possible Relevance of Soluble Luteinizing Hormone Receptor during Development and Adulthood in Boys and Men. Cancers (Basel). 2021 Mar 16;13(6):1329. doi: 10.3390/cancers13061329. PMID 33809538